CLINICAL TRIAL: NCT00484640
Title: Modeling Genotype and Other Factors to Enhance the Safety of Coumadin Prescribing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Collaborators: Marshfield Clinic Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01HS016335-01 (AHRQ)
Record Dates: First submitted 2007-06-04; First posted 2007-06-11 (Estimated); Last update posted 2007-06-11 (Estimated); Status verified 2007-06

CONDITIONS: Atrial Fibrillation; Deep Venous Thrombosis; Heart Valve Replacement; Pulmonary Embolism
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Coumadin

SUMMARY:
The study goal is to conduct a randomized controlled trial to compare safety and accuracy of dosing based on clinical information including the clinical reason for your taking coumadin, your age, gender, your body surface area, and other medical conditions you may have with dosing estimated by a dosing calculator which adjusts for factors affecting coumadin dosing variability including genotypes for genes important in Coumadin metabolism and response. The hypothesis to be tested by this trial states that:when compared to patients managed with a best practices standard-of-care coumadin dosing regimen, patients randomized to coumadin dosing based on genetically programmed metabolic capacity and other known clinical and environmental factors affecting dose will: 1)show reduced risk of adverse events (using surrogate measures of such events); and 2)more rapidly achieve Coumadin dosing.

DETAILED DESCRIPTION:
The study goal is to conduct a randomized controlled trial to compare safety and accuracy of dosing based on clinical information including clinical reason for taking coumadin, your age, gender, your body surface area, and other medical conditions you may have and dosing with dosing estimated by a dosing calculator which adjusts for factors affecting coumadin dosing variability including genotypes for genes important in Coumadin metabolism and response. The hypothesis to be tested by this trial states that:when compared to patients managed with a best practices standard-of-care coumadin dosing regimen, patients randomized to coumadin dosing based on genetically programmed metabolic capacity and other known clinical and environmental factors affecting dose will: 1)show reduced risk of adverse events (using surrogate measures of such events); and 2)more rapidly achieve Coumadin dosing

ELIGIBILITY:
Inclusion Criteria:

* Caucasian male and female patients(including Hispanic white) greater than or equal to 40 years of age;
* Patients initiating coumadin therapy without a documented history of stabilized dose of coumadin therapy;
* Target INR of 2 to 3.5;
* Women of childbearing potential must use an effective method of birth control(e.g. condom,oral contraceptives, indwelling intrauterine device, abstinence.

Exclusion Criteria:

* Age less than 40 years;
* Patients of known Native American, Asian, or African descent;
* Patients with thrombocytopenia(platelet count<50x10 cells/ml);
* Patient has previously received coumadin and information on dosing of the patient is known at time of restarting coumadin;
* Patients with severe to moderate hepatic insufficiency (AST or ALT less than 2x the upper limit of normal;
* Clinical contraindication for coumadin therapy;
* Female patients with a positive pregnancy test or women who are breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2007-06; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
weighted time in therapeutic range
absolute deviation from clinically optimal dose

SECONDARY OUTCOMES:
time to stable dose in therapeutic target range
warfarin related adverse drug events
time to first INR above 4

CONTACTS AND LOCATIONS:
Overall Officials: Michael Caldwell, Physician, Principal Investigator — Marshfield Clinic Research Foundation
Locations (2):
- United States (2):
  - Third Wave Molecular Diagnostics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin

REFERENCES:
- [Background] Hillman MA, Wilke RA, Caldwell MD, Berg RL, Glurich I, Burmester JK. Relative impact of covariates in prescribing warfarin according to CYP2C9 genotype. Pharmacogenetics. 2004 Aug;14(8):539-47. doi: 10.1097/01.fpc.0000114760.08559.dc. PMID 15284536
- [Background] Greenlee RT, Vidaillet H. Recent progress in the epidemiology of atrial fibrillation. Curr Opin Cardiol. 2005 Jan;20(1):7-14. PMID 15596953
- [Background] Wilke RA, Berg RL, Vidaillet HJ, Caldwell MD, Burmester JK, Hillman MA. Impact of age, CYP2C9 genotype and concomitant medication on the rate of rise for prothrombin time during the first 30 days of warfarin therapy. Clin Med Res. 2005 Nov;3(4):207-13. doi: 10.3121/cmr.3.4.207. PMID 16303885
- [Background] Hillman MA, Wilke RA, Yale SH, Vidaillet HJ, Caldwell MD, Glurich I, Berg RL, Schmelzer J, Burmester JK. A prospective, randomized pilot trial of model-based warfarin dose initiation using CYP2C9 genotype and clinical data. Clin Med Res. 2005 Aug;3(3):137-45. doi: 10.3121/cmr.3.3.137. PMID 16160068